CLINICAL TRIAL: NCT00188786
Title: A Phase II Feasibility Study of Cone Beam Computed Tomography for Daily Image Guidance in Patients Receiving Dose Escalated Conformal Radiation Therapy for Prostate Cancer
Brief Title: Cone Beam CT for Daily Image Guidance - Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Dr Charles Catton, Staff Radiation Oncologist, University Health Network, Princess Margaret Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 05-0037-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: daily Cone Beam CT for imaging guidance for radiotherapy

SUMMARY:
Conformal dose escalated radiation therapy (CRT) is standard treatment for patients with low and intermediate risk prostate cancer. CRT requires accurate daily localization of the prostate prior to treatment to correct for prostate motion and set-up errors. Cone beam computed tomography (CT) can accurately localize fiducial markers within the prostate. Cone Beam CT also provides important information on daily position of organs within the pelvis. This study aims to assess the feasibility of cone beam CT for daily localization of the prostate as well as document changes in size and location of pelvic organs during an entire course of CRT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate
* Patient undergoing dose escalated conformal external beam radiation therapy
* Low or intermediate risk prognostic factors (PSA 20 or less, Gleason score <8, Clinical T category <T3, Clinical N category 0 or X, M category 0 or X
* Age 18 years or older
* ECOG performance status 0 or 1
* Informed consent

Exclusion Criteria:

* Inflammatory bowel disease or collagen vascular disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of cone beam CT for daily on-line image guidance in patients receiving conformal radiation therapy for prostate cancer.

SECONDARY OUTCOMES:
To measure the amount of interfraction movement of the prostate and seminal vesicles with current bowel regimen of daily milk of magnesia.
To measure the amount of interfraction movement and deformity of the rectum and bladder with current bowel regimen of daily milk of magnesia.
To develop a technique for delivery of radiation therapy that reduces normal tissue toxicity, based on rectal and bladder avoidance models.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Catton, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada